CLINICAL TRIAL: NCT00248898
Title: Quality of Life After Open Heart Surgery in Older Patients
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0501007700
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Open Heart Surgery Patients
Keywords: nonagenarians; quality of life; cardiothoracic surgery; long term survival
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac Surgery — Coronary artery bypass graft surgery, aortic valve replacement, mitral valve replacement, aortic aneurysm repair

SUMMARY:
Long term follow-up of nonagenarians who have undergone open heart procedures.

DETAILED DESCRIPTION:
Based on population studies, life expectancy at age 80 is 8.5 years, and at the age of 85 years, it is 6.3 years (US Bureau of Census 2000). There are currently 1.6 million nonagenarians and roughly 72,000 centenarians living in the United States. With this increasing elderly population, knowledge of the special management issues and long-term sequela are imperative. Bacchetta and coworkers from our institution presented a 10-year outcomes experience in nonagenarians undergoing cardiac surgery. In 42 consecutive patients, in-hospital mortality was 7%, and 30-day mortality 5%. Postoperative morbidity was documented in 67% with arrhythmias accounting for 31% of the cases, followed by respiratory complications, infections, and strokes. While this is mostly in-hospital data, long-term follow-ups have not been performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent open heart procedures and who were 90 years or greater between 1995 and 2004 at The New York Presbyterian Hospital

Exclusion Criteria:

* Patients who refuse follow-up

Min Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A (consecutive) series of 49 patients age 90 years or older underwent cardiac operations between May 1995 and October 2004 at New York Presbyterian Hospital-Weill Medical College of Cornell University.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl H Krieger, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital - Weill Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators may contact the PI for access to the data, with their planned analyses

REFERENCES:
- [Background] Ullery BW, Peterson JC, Milla F, Wells MT, Briggs W, Girardi LN, Ko W, Tortolani AJ, Isom OW, Krieger KH. Cardiac surgery in select nonagenarians: should we or shouldn't we? Ann Thorac Surg. 2008 Mar;85(3):854-60. doi: 10.1016/j.athoracsur.2007.10.074. PMID 18291156